CLINICAL TRIAL: NCT05295043
Title: A Multicenter Clinical Study Evaluating Real-world CDK4/6 Inhibitor Combined With Endocrine Therapy in HR+/HER2- Advanced Breast Cancer
Brief Title: Advanced Breast Cancer Study of CDK4/6 Inhibitor Combined With Endocrine Therapy Endocrine Therapy in HR+/HER2- Advanced Breast Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: BC-RWS
Record Dates: First submitted 2022-03-15; First posted 2022-03-24 (Actual); Last update posted 2022-09-29 (Actual); Status verified 2022-03

CONDITIONS: Advanced HR+ HER2 Negative Breast Carcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HR+/HER2- advanced breast cancer patients receiving CDK4/6 inhibitor combined with endocrine therapy (Experimental): According to clinical guidelines or drug instructions, the treating physician will adjust the drug dose in accordance with the clinical reality and the patient's personal situation.
  Interventions: Drug: (CDK)4/6 inhibitor

INTERVENTIONS:
Drug: (CDK)4/6 inhibitor — CDK4/6 inhibitor + AI/fulvestrant therapy，According to clinical guidelines or drug instructions, the treating physician will adjust the drug dose in accordance with the clinical reality and the patient's personal situation.
  Other Names: ET

SUMMARY:
By retrospectively collecting and arranging real-world data of multi-center HR+/HER2- advanced breast cancer in China combined with CDK4/6 inhibitor and endocrine therapy, we analyzed different HER2 expression levels (HER2 0, 1+, 2+ and FISH-), especially Clinical outcomes of endocrine therapy for metastatic breast cancer with low HER2 expression (HER2 1+, 2+ and FISH-), exploring potential biomarkers of CDK4/6 inhibitors, and understanding the outcome characteristics of HER2 heterogeneity in MBC through multivariate analysis , and guide clinical application.

ELIGIBILITY:
Inclusion Criteria:

* 1) Female patients with advanced breast cancer aged ≥18 years. 2) For breast cancer patients diagnosed as HR-positive and HER2-negative by pathological examination, the expression levels of ER, PR, and HER2 were reported by immunohistochemistry in the primary or metastatic lesions.

  1. ER positivity and/or PR positivity is defined as: the proportion of tumor cells with positive staining accounts for ≥ 10% of all tumor cells (confirmed by the investigator of the trial center);
  2. HER2 negative is defined as: standard immunohistochemistry (IHC) test is 0/1+; HER2 (2+) needs to be tested by FISH, HER2/CEP17 ratio is less than 2.0 or HER2 gene copy number is less than 4 (by the test center of the test center) Investigator review and confirmation).

     3) CDK4/6 inhibitors combined with endocrine therapy can conduct complete efficacy evaluation and follow-up information collection.

     4) Postmenopausal or premenopausal/perimenopausal female patients can be enrolled.

     Postmenopausal status, defined as meeting at least one of the following criteria: prior bilateral ovarian surgery; age ≥60 years; age <60 years, menopause for at least 12 months (not due to chemotherapy, tamoxifen, toremide) fen or ovarian suppression) and follicle-stimulating hormone (FSH) and estrogen levels are in the postmenopausal range.

     Premenopausal or perimenopausal women may also be enrolled, but must be willing to receive LHRHa during the study period.

     5) According to RECIST 1.1 criteria, patients must have: a) measurable lesions; b) unmeasurable osteolytic or mixed (osteolytic + osteoblastic) bone lesions in the absence of measurable lesions.

     Exclusion Criteria:
* 1) Early breast cancer patients receive CDK4/6 inhibitor drug therapy. 2) HER2 overexpression or gene amplification, such as immunohistochemical score 3+ or positive fluorescence in situ hybridization.

  3) Pregnant or lactating female patients. 4) Patients deemed unsuitable for inclusion by the investigator.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2022-12-10 (Estimated); Primary Completion 2024-01-01 (Estimated); Study Completion 2024-01-01 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) From enrollment to progression or death (for any reason) Progression-free survival (PFS) | Estimated 24 months
  From enrollment to progression or death (for any reason)

SECONDARY OUTCOMES:
Objective response rate (ORR) | Estimated 24 months
  Ratio of CR and PR in all subjects
Disease Control Rate (DCR) | Estimated 24 months
  Ratio of CR ,PR and SD in all subjects
Overall survival (OS) | Estimated 36 months
  From enrollment to death (for any reason)